CLINICAL TRIAL: NCT02689960
Title: Vaginal Prednisone Administration for Prevention of Adrenal Crisis - a Bioequivalence Study
Brief Title: Vaginal Prednisone Administration for Prevention of Adrenal Crisis
Acronym: Vapreda
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Vapreda
Record Dates: First submitted 2016-02-08; First posted 2016-02-24 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-05

CONDITIONS: Adrenal Insufficiency
Keywords: addison disease; adrenal crisis; prednisone
MeSH Terms: conditions — Adrenal Insufficiency; Addison Disease | interventions — Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vaginal administration first (Other): Intervention first visit: vaginal administration of 100mg prednisone suppository, Intervention second visit: rectal administration of 100mg prednisone suppository
  Interventions: Drug: 100mg prednisone suppository
- rectal administration first (Other): Intervention first visit: rectal administration of 100mg prednisone suppository, Intervention second visit: vaginal administration 100mg prednisone suppository
  Interventions: Drug: 100mg prednisone suppository

INTERVENTIONS:
Drug: 100mg prednisone suppository — vaginal administration of 100mg prednisone suppository (Rectodelt)
  Other Names: Rectodelt (approval number 6329964.00.00)

SUMMARY:
Patients with chronic adrenal insufficiency need to adapt their glucocorticoid replacement dose in conditions of physical or psychological stress to prevent life threatening adrenal crisis. In cases of more severe impairment or unsecure gastrointestinal absorption (e.g. gastroenteritis, severe infectious disease), rapid and highly dosed administration of glucocorticoids is crucial. The study is conducted to offer female patients the possibility to perform efficient prednisone self-administration in emergency situations in a way of administration, which is easy to perform and accepted by the patients. Therefore, pharmacokinetics and safety of vaginal prednisone administration will be studied and compared to rectal administration.

DETAILED DESCRIPTION:
As patients with adrenal insufficiency still die from adrenal crisis, improvement of both prevention and also emergency management is needed. It is clear that perfect equipment and education of patients is key for further crisis prevention and management. Vaginal administration of prednisone-suppositories is easy to perform and independent of the gastro-intestinal system. Thus, this study aims at the efficacy, feasibility and safety of vaginal administration of prednisone-suppositories.

Recruitment:

Patients with primary adrenal insufficiency will be recruited. The adrenal insufficiency registry of Würzburg comprises more than 150 patients with primary adrenal insufficiency. Several patients have already indicated their interest to participate in the study. According to the European Medicines Agency (EMA) notes for guidance on the investigation of bioavailability and bioequivalence the number of 12 participants is regarded as the minimum required number.

Trial flow:

Pharmacokinetic studies will be performed at two different study visits. Patients will receive a 100mg prednisone suppository (Rectodelt® 100 mg) vaginal and rectal on two different study visits (interval longer then one week). Blood samples for determination of prednisone and adrenocorticotropic Hormone (ACTH) levels will be collected over a time period of 6 hours. Patients receive a diary to document eventual local or systemic adverse events during the following 7 days.

Stopping rules:

Participation of patients is fully voluntarily. Patients are able to stop participation in the study at any point in time. In addition, patients might claim the elimination of all data material at any point in time. Furthermore, study participation will be stopped for the individual patient, if new safety issues occur (e. g. new diagnosis of Diabetes mellitus, pregnancy or acute infectious disease) during the study. Relevant risks to the patients are highly unlikely. However, if 2 or more patients experience serious adverse events associated with the vaginal administration of prednisone with high likelihood, the study will be stopped.

Written informed consent:

A consent document including patient information upon the nature, scope and possible consequence of the trial must have been approved by the Institutional Review Board. Patients amenable for inclusion in the trial will be given sufficient time to study the written information, as well as possibility to ask questions before signing the consent document.

Analysis:

Documentation and analysis will be performed at the Department of Medicine I, Endocrine and Diabetes Unit, University of Würzburg, Germany. Data will be documented after pseudonymisation in a data base. Data analysis is mainly descriptive (bioequivalence of vaginal prednisone administration compared to rectal application, estimation of the patients regarding convenience and tolerability of different modes of drug administration, safety aspects).

Safety:

In the course of the trial, changes in physical findings as well as clinical signs and symptoms that may reflect adverse effects will be documented. Furthermore, all adverse events will be documented on the appropriate report form. When an adverse event occurs it will be graded according to the National cancer Institute - common toxicity criteria (NCI-CTC) (version 4.0). Patients receive a diary to document any local or systemic adverse event during the following 7 days after intervention. In addition, patients will be contacted by phone 3(±1) and 7(±1) days after vaginal administration of prednisone. If patients report any adverse events that are possibly related to the vaginal administration route, they will be called-in for further physical examination and detailed documentation. To further enhance individual patient's safety during the study, a safety assessment will be performed prior to the subsequent intervention. In addition, a safety assessment will be performed after 4 and 8 subsequent vaginal administrations of prednisone with evaluation of events during the 7 day follow up period after administration.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with chronic primary adrenal insufficiency due to autoimmune adrenalitis or bilateral adrenalectomy (disease duration at least 6 months)
* Age ≥ 18 years
* Patient´s written informed consent
* Ability to comply with the protocol procedures
* Established stable replacement therapy, no anticipated change in medication
* Negative pregnancy test and contraception (besides oral contraceptive pill) in pre-menopausal females

Exclusion Criteria:

* Diabetes mellitus
* Infectious disease with fever at time of investigation
* Known intolerance to the study drug or constituents
* Oral contraception
* Pregnancy or breast feeding
* Renal failure (creatinine >2.5 ULN)
* Disposition to vaginal mycosis (requiring treatment in the last 6 months or of necessity >2 antimycotic therapies/year)
* Recurrent urinary tract infections (of necessity >2 antibiosis therapies/year)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Bioequivalence of vaginal prednisone administration compared to rectal application, assessed by repeated determination of prednisolon levels (in blood) | up to 12 months
  The hypothesis is that the same prednisolone levels can be achieved within the same time frame after vaginale administration compared to rectal application.

SECONDARY OUTCOMES:
Safety of the vaginal administration of prednisone compared to rectal application, assessed by the number of participants with treatment-related adverse events (using the NCI-CTC, version 4.0). | up to 12 months
Suppressive effects on ACTH levels after vaginal administration of prednisone compared to rectal application, assessed by repeated determination of ACTH-levels | up to 1 week
  ACTH-levels are measured in plasma
Tolerability by the patients assessed by a questionnaire | up to 1 month
  Questions record the preference of the patients between vaginal and rectal application.

CONTACTS AND LOCATIONS:
Overall Officials: Stefanie Hahner, MD, Prof., Principal Investigator — University Hospital Wuerzburg

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Hahner S, Spinnler C, Fassnacht M, Burger-Stritt S, Lang K, Milovanovic D, Beuschlein F, Willenberg HS, Quinkler M, Allolio B. High incidence of adrenal crisis in educated patients with chronic adrenal insufficiency: a prospective study. J Clin Endocrinol Metab. 2015 Feb;100(2):407-16. doi: 10.1210/jc.2014-3191. Epub 2014 Nov 24. PMID 25419882
- [Background] Hahner S, Hemmelmann N, Quinkler M, Beuschlein F, Spinnler C, Allolio B. Timelines in the management of adrenal crisis - targets, limits and reality. Clin Endocrinol (Oxf). 2015 Apr;82(4):497-502. doi: 10.1111/cen.12609. Epub 2014 Nov 6. PMID 25200922
- [Background] Hahner S, Loeffler M, Bleicken B, Drechsler C, Milovanovic D, Fassnacht M, Ventz M, Quinkler M, Allolio B. Epidemiology of adrenal crisis in chronic adrenal insufficiency: the need for new prevention strategies. Eur J Endocrinol. 2010 Mar;162(3):597-602. doi: 10.1530/EJE-09-0884. Epub 2009 Dec 2. PMID 19955259
- [Background] Hahner S, Burger-Stritt S, Allolio B. Subcutaneous hydrocortisone administration for emergency use in adrenal insufficiency. Eur J Endocrinol. 2013 Jun 29;169(2):147-54. doi: 10.1530/EJE-12-1057. Print 2013 Aug. PMID 23672956
- [Background] Allolio B. Extensive expertise in endocrinology. Adrenal crisis. Eur J Endocrinol. 2015 Mar;172(3):R115-24. doi: 10.1530/EJE-14-0824. Epub 2014 Oct 6. PMID 25288693
- [Background] Smans LC, Van der Valk ES, Hermus AR, Zelissen PM. Incidence of adrenal crisis in patients with adrenal insufficiency. Clin Endocrinol (Oxf). 2016 Jan;84(1):17-22. doi: 10.1111/cen.12865. Epub 2015 Aug 27. PMID 26208266
- [Background] Anderson M, Kutzner S, Kaufman RH. Treatment of vulvovaginal lichen planus with vaginal hydrocortisone suppositories. Obstet Gynecol. 2002 Aug;100(2):359-62. doi: 10.1016/s0029-7844(02)02117-8. PMID 12151163